CLINICAL TRIAL: NCT07327372
Title: Effect of Perineural Dexmedetomidine as an Adjuvant to Pericapsular Nerve Group Block in Older Adults: A Randomized Controlled Trial
Brief Title: PENG Block With Dexmedetomidine in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16/2025
Record Dates: First submitted 2025-12-28; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hip Osteoarthritis; Arthropathy of Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Ropivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG Block With Ropivacaine (Active Comparator): Participants will receive an ultrasound-guided pericapsular nerve group (PENG) block using ropivacaine 0.2%, total volume 20 mL, administered as a single perineural injection prior to surgery. The block will be performed according to a standardized protocol by an experienced anesthesiologist.
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- PENG Block With Ropivacaine Plus Dexmedetomidine (Experimental): Participants will receive an ultrasound-guided pericapsular nerve group (PENG) block using ropivacaine 0.2% (20 mL) combined with dexmedetomidine 25 micrograms, administered as a single perineural injection prior to surgery. The block will be performed according to a standardized protocol by an experienced anesthesiologist.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — Ropivacaine is a long-acting local anesthetic used for regional anesthesia. In this study, it is administered perineurally as part of an ultrasound-guided pericapsular nerve group (PENG) block for postoperative pain management in older adults undergoing hip surgery.
  Other Names: Ropivacaine hydrochloride
  Arms: PENG Block With Ropivacaine
Drug: Dexmedetomidine — Dexmedetomidine is a selective alpha-2 adrenergic agonist used as an adjuvant to local anesthetics to enhance and prolong analgesia. In this study, dexmedetomidine is administered perineurally in combination with ropivacaine as part of an ultrasound-guided pericapsular nerve group (PENG) block.
  Other Names: Dexmedetomidine hydrochloride
  Arms: PENG Block With Ropivacaine Plus Dexmedetomidine

SUMMARY:
Pain after hip surgery is a common problem in older adults and may delay early mobilization, increase the need for opioid pain medications, and contribute to complications such as delirium, nausea, or prolonged hospital stay. Regional anesthesia techniques are increasingly used to improve pain control while reducing the use of systemic opioids.

The pericapsular nerve group (PENG) block is a modern ultrasound-guided regional anesthesia technique designed to provide effective pain relief after hip surgery while preserving muscle strength. It allows patients to begin mobilization earlier and may reduce the risk of postoperative complications, which is particularly important in older adults.

Ropivacaine is a commonly used local anesthetic for nerve blocks. Dexmedetomidine is a medication that, when added in small doses to local anesthetics, may prolong pain relief and improve the quality of nerve blocks without significantly increasing side effects. However, the benefits and safety of adding dexmedetomidine to the PENG block in older adults have not been sufficiently studied.

The aim of this randomized controlled clinical study is to compare the effectiveness and safety of two PENG block techniques in older adults undergoing hip surgery. Participants will be randomly assigned to one of two groups. One group will receive a PENG block with 20 mL of 0.2% ropivacaine. The second group will receive a PENG block with 20 mL of 0.2% ropivacaine combined with 25 micrograms of dexmedetomidine.

The study hypothesis is that the addition of dexmedetomidine to ropivacaine in the PENG block will provide longer-lasting and more effective postoperative pain relief compared with ropivacaine alone, without increasing adverse effects. Outcomes assessed in the study will include postoperative pain intensity, need for additional pain medications, time to first mobilization, and the occurrence of side effects such as low blood pressure, slow heart rate, excessive sedation, or delirium.

The results of this study may help optimize regional anesthesia techniques for hip surgery in older adults and contribute to safer, more effective postoperative pain management strategies.

DETAILED DESCRIPTION:
Postoperative pain following hip surgery is a significant clinical problem in older adults and is associated with delayed mobilization, increased opioid consumption, higher risk of delirium, and prolonged hospitalization. Effective pain control that preserves motor function is particularly important in this population to support early rehabilitation and reduce postoperative complications.

The pericapsular nerve group (PENG) block is an ultrasound-guided regional anesthesia technique that targets the sensory innervation of the anterior hip capsule while sparing motor nerves. This technique has been shown to provide effective analgesia after hip surgery and may facilitate early postoperative mobilization. However, the duration of analgesia achieved with local anesthetics alone may be limited.

Ropivacaine is a long-acting local anesthetic commonly used for peripheral nerve blocks. Dexmedetomidine is an alpha-2 adrenergic agonist that has been used as an adjuvant to local anesthetics to prolong analgesia and improve block quality. When administered in low perineural doses, dexmedetomidine may enhance analgesic duration without causing clinically significant systemic side effects. Nevertheless, data regarding its use as an adjuvant to the PENG block in older adults are limited.

This study is designed as a prospective, randomized, controlled clinical trial comparing two PENG block regimens in older adults undergoing hip surgery. Eligible participants will be randomly assigned to one of two groups. The control group will receive a PENG block with 20 mL of 0.2% ropivacaine. The intervention group will receive a PENG block with 20 mL of 0.2% ropivacaine combined with 25 micrograms of dexmedetomidine. The PENG block will be performed under ultrasound guidance by experienced anesthesiologists according to a standardized protocol.

All participants will receive standardized general or regional anesthesia for surgery and postoperative multimodal analgesia according to institutional protocols. Postoperative pain management will be identical in both groups, except for the study intervention, to minimize confounding factors.

The primary objective of the study is to assess whether the addition of dexmedetomidine to ropivacaine prolongs and improves postoperative analgesia provided by the PENG block compared with ropivacaine alone. Secondary objectives include evaluation of postoperative pain intensity, total opioid consumption, time to first mobilization, and patient comfort.

Safety outcomes will also be assessed, with particular attention to adverse effects relevant to older adults, including hypotension, bradycardia, excessive sedation, nausea, vomiting, and postoperative delirium. Hemodynamic parameters and sedation levels will be monitored routinely in the postoperative period.

The results of this study are expected to provide clinically relevant information on the efficacy and safety of dexmedetomidine as an adjuvant to the PENG block in older adults. These findings may contribute to the optimization of regional anesthesia strategies and improved postoperative pain management in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Scheduled for elective or emergency hip surgery (e.g., hip fracture fixation or hip arthroplasty)
* ASA physical status I-III
* Ability to communicate pain intensity using the NRS scale
* Written informed consent obtained from the patient or legal representative
* Planned use of PENG block as part of multimodal perioperative analgesia

Exclusion Criteria:

* Patient refusal or inability to provide informed consent
* Allergy, intolerance, or contraindication to any study medication: ropivacaine, dexmedetomidine
* Pre-existing neurological deficit or neuropathy of the affected limb
* Coagulopathy (INR >1.5, platelets <100,000/µL) or current therapeutic anticoagulation that contraindicates regional anesthesia
* Infection at or near the injection site
* Severe hepatic or renal impairment
* History of chronic opioid use (daily opioids >30 days before surgery)
* Cognitive impairment or delirium precluding reliable pain assessment
* BMI > 40 kg/m² (if you want to exclude for technical difficulty)
* Patients receiving another regional nerve block for hip surgery
* Pregnancy or breastfeeding
* Participation in another interventional clinical trial within 30 days

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to First Rescue Analgesia | Within 48 hours after the end of surgery
  Time (in hours) from the end of the PENG block (completion of local anesthetic injection) to the first administration of rescue analgesia (opioid or non-opioid) given for pain intensity ≥4 on the 0-10 Numerical Rating Scale (NRS). Data will be collected from anesthesia records and postoperative medication charts.

SECONDARY OUTCOMES:
Pain Intensity at Rest (NRS 0-10) | 4 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 8 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 12 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 24 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 48 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 4 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 8 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 12 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 24 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 48 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Total Opioid Consumption | 0-48 hours after surgery
  Cumulative dose of all opioid analgesics administered in the postoperative period, converted to oral morphine milligram equivalents (MME). Values at 24 and 48 hours will be recorded and compared between groups.
Block-Related Adverse Events, Including Neurological Complications | From block placement until hospital discharge, up to 30 days
  Incidence of complications potentially related to the PENG block or perineural adjuvants, including signs of local anesthetic systemic toxicity, prolonged motor or sensory deficit, nerve injury (evaluated in the postoperative clinic or outpatient nerve injury clinic if required), infection at the injection site, hematoma, or persistent weakness.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, MD PhD, Study Chair — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after publication
Access Criteria: Upon reasonable request